CLINICAL TRIAL: NCT02737553
Title: Enclosed Electromechanical Morcellation and Vaginal Removal During Laparoscopic Myomectomy
Brief Title: Laparoscopic Enclosed Morcellation; Electromechanic Morcellation vs Vaginal Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ali Akdemir, Ali Akdemir MD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAkdemir1
Record Dates: First submitted 2016-03-21; First posted 2016-04-14 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-02

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enclosed morcellation (Active Comparator): In this group, after extirpation of the myoma from the uterus and repair of the uterine defect, the myoma will be removed from the abdomen with an enclosed laparoscopic electromechanical morcellation as described in the literature by Akdemir et al with using surgical glove (Akdemir A et. al, Innovative technique for enclosed morcellation using a surgical glove. Obstet Gynecol. 2015 May;125(5):1145-9.
  doi: 10.1097/AOG.0000000000000823.).
  Interventions: Procedure: Enclosed morcellation
- vaginal morcellation (Active Comparator): In this group, after extirpation of myoma from uterus and repair of the uterine defect, myoma will be removed through the vagina with posterior colpotomy. In this group myoma will also be removed in a enclosed fashion with using endo bag.
  Interventions: Procedure: vaginal morcellation

INTERVENTIONS:
Procedure: Enclosed morcellation — After extirpation of the myoma from the uterus and repair of the uterine defect, the myoma will be removed from the abdomen with an enclosed laparoscopic electromechanical morcellation as described in the literature by Akdemir et al with using surgical glove (Akdemir A et. al, Innovative technique for enclosed morcellation using a surgical glove. Obstet Gynecol. 2015 May;125(5):1145-9. doi: 10.1097/AOG.0000000000000823.).
  Arms: enclosed morcellation
Procedure: vaginal morcellation — After extirpation of myoma from uterus and repair of the uterine defect, myoma will be removed through the vagina with posterior colpotomy. In this group myoma will also be removed in a enclosed fashion with using endo bag.
  Arms: vaginal morcellation

SUMMARY:
Laparoscopic tissue removal is one of the most challenging parts for the laparoscopic surgery. For this reason, electromechanical morcellation has long been used to facilitate the tissue removal in gynecology. However, electromechanical morcellation has long been performed inside the abdomen without any containment. Therefore, this practice has recently undergone increased scrutiny because of important concerns related to tissue dissemination during intracorporeal power morcellation. Thus, the US Food and Drug Administration released a safety communication discouraging power morcellation in laparoscopic hysterectomy and myomectomy procedures in April 2014.

As a result of this serious concern, the enclosed laparoscopic power morcellation has been come into prominence in gynecological surgery. Besides the removal of the tissues through vagina with posterior colpotomy is considered an another solution for this critical problem.

In the literature the comparison for the two techniques for tissue removal is considerably scarce. Therefore researchers are aiming to prepare a trial to compare the laparoscopic enclosed electromechanical morcellation and tissue removal thorough vagina with posterior colpotomy according to surgical time, postoperative pain and postoperative sexual function.

DETAILED DESCRIPTION:
In this study researchers aiming to compare the compare the laparoscopic enclosed electromechanical morcellation and tissue removal thorough vagina with posterior colpotomy according to surgical time, postoperative pain and postoperative sexual function.

Patients with an indication of myomectomy, between 18 to 40 years old, without prior abdominal surgery and without suspicious of malignancy will include into the study. Anticipated number of the patients will be 60. Participants will be randomized into two groups; group 1 enclosed electromechanical morcellation will be performed to remove the myoma out of the abdominal cavity; group 2 myoma will be removed through vagina with posterior colpotomy. In group 1, after extirpation of the myoma from the uterus and repair of the uterine defect, the myoma will be removed from the abdomen with an enclosed laparoscopic electromechanical morcellation with using surgical glove. In group 2, after extirpation of myoma from uterus and repair of the uterine defect, myoma will be removed through the vagina with posterior colpotomy. In this group myoma will also be removed in a enclosed fashion with using endo bag. Tissue removal time (for group 1 removal time is decided time between the insertion and removal of the morcellation, for group two removal time is decided time between start of the posterior colpotomy and end of the closure of the posterior colpotomy), postoperative time and sexual function of the patient and any of the complications will be compared. Visual pain score and female sexual function index questionnaire will be used to assess the postoperative pain and sexual function, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Myoma Uteri
* No prior abdominal surgery

Exclusion Criteria:

* Suspicious for malignancy
* Prior abdominal surgery
* no vaginal intercourse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akdemir, MD, Principal Investigator — Ege University
Locations (1):
- Department of Obstetrics and Gynecology, Ege University School of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen patients with prior abdominal surgery and 4 participants without previous vaginal intercourse were excluded from the study.
Groups:
- Enclosed Morcellation: In this group, after extirpation of the myoma from the uterus and repair of the uterine defect, the myoma will be removed from the abdomen with an enclosed laparoscopic electromechanical morcellation as described in the literature by Akdemir et al with using surgical glove.
- Vaginal Morcellation: In this group, after extirpation of myoma from uterus and repair of the uterine defect, myoma will be removed through the vagina with posterior colpotomy.
Period: Overall Study
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
Started | 49 | 48
Completed | 49 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enclosed Morcellation | Vaginal Morcellation | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (5.9) | 35.5 (3.2) | 36.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (2.9) | 26.6 (5.2) | 25.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Operation Time
Description: Total operation time will be compared between two groups in seconds.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
Number analyzed (Participants) | 49 | 48
seconds | 146.1 (31.6) | 124.6 (35.4)

2. Secondary Outcome: Morcellation Time
Description: After extirpation of the myoma in group 1 the fibroid was placed into the glove within the abdomen. The morcellation was accomplished within the completely enclosed glove. In Group 2, after extirpation of the myoma, it was removed through the vagina through posterior colpotomy. An endoscopic specimen bag was placed into the abdomen following the vaginal posterior colpotomy. Then, the fibroid was placed into the endoscopic bag within the abdomen. The specimen was removed with coring technique via scalpel. Posterior colpotomy incision was then sutured vaginally.
  Morcellation time is decided time between the insertion and removal of the surgical glove in group 1 and time between start of the posterior colpotomy and end of the closure of the posterior colpotomy in group 2. Tissue morcellation time compared between two groups in seconds.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
Number analyzed (Participants) | 49 | 48
seconds | 25.94 (8.1) | 20.79 (6.9)

3. Other Pre Specified Outcome: Postoperative Pain
Description: Postoperative pain was compared between two groups using visual analog score in 0 to 10 scale.
  Participants were assessed in terms of pain with the Visual Pain Scale (VAS). The participants were asked to rate current pain on a 10-cm visual analog scale (VAS), with 0 being no pain and 10 the worst pain imaginable 48 hours after operation.
Time Frame: 2 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Enclosed Morcellation: In this group, after extirpation of the myoma from the uterus and repair of the uterine defect, the myoma will be removed from the abdomen with an enclosed laparoscopic electromechanical morcellation as described in the literature.
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
Number analyzed (Participants) | 49 | 48
score on a scale | 1.7 (1.6) | 1.6 (1.38)

4. Other Pre Specified Outcome: Sexual Functional Assessment
Description: Sexual function will be assessed with using "Female Sexual Function Index questionnaire" and it will be compared between two groups.
  Participants were requested to fill FSFI (Female Sexual Function Index) forms to evaluate their sexual lives. The FSFI consists of 19 questions and is a validated questionnaire for the assessment of sexual function. The questions are grouped into the subdomains of libido, arousal, lubrication, orgasm, satisfaction, and pain. The total score is determined by summing up the subdomains scores. Higher scores reflect better sexual function; maximum score is 36 and minimum score is 0. For each subdomain, higher scores reflect better sexual function; maximum score is 6 and minimum score is 0 including pain, in which 0 reflects lots of pain and 6 reflects the absence of pain.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
Number analyzed (Participants) | 49 | 48
score on a scale | 18.4 (9.9) | 25.3 (4.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Enclosed Morcellation | Vaginal Morcellation
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT02737553/Prot_SAP_000.pdf